CLINICAL TRIAL: NCT04539925
Title: Impact of Short-term Air Pollution Exposure on Acute Coronary Syndrome in Two Cohorts of Industrial and Non-industrial Areas: A Time Series Regression With 6,000,000 Person-years of Follow-up (ACS - Air Pollution Study)
Brief Title: Air Pollution Exposure on Acute Coronary Syndrome in Two Cohorts of Industrial and Non-industrial Areas
Status: Completed | Type: Observational
Sponsor: Medical University of Silesia (Other)
Collaborators: Medical University of Bialystok (Other)
Responsible Party: Principal Investigator, Wojciech Wańha, MD, PhD, Medical University of Silesia
Other Study IDs: 03
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-08

CONDITIONS: Acute Coronary Syndrome; Air Pollution
Keywords: Acute Coronary Syndrome; Air pollution
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Industrial area
  Interventions: Other: Acute coronary syndrome
- Non-industrial area
  Interventions: Other: Acute coronary syndrome

INTERVENTIONS:
Other: Acute coronary syndrome — The effect of air pollution on acute coronary syndrome

SUMMARY:
Background: There is a lack of data on the effect of air pollution on acute coronary syndrome (ACS) in industrial and non-industrial areas.

Objectives: A comparison of association of air pollution exposure with ACS in two cohorts of industrially different areas.

Materials and methods: The study covered 6,000,000 person-years of follow-up and five types of air pollution between 2008 and 2017. A time series regression analysis with 7-lag was used to assess the effects air pollution on ACS.

ELIGIBILITY:
The study covered all residents from industrial (Katowice) and non-industrial (Białystok) areas.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study is performed in two big provincial cities in Poland, Europe, namely Bialystok and Katowice. In the last year of the analysis, the areas were inhabited by 294,925 and 296,262 residents, respectively.
Sampling Method: Probability Sample
Enrollment: 9046 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Non-ST segment elevation myocardial infarction | 7 days
ST-segment elevation myocardial infarction | 7 days

CONTACTS AND LOCATIONS:
Locations (2):
- Poland (2):
  - Department of Invasive Cardiology, Medical University of Bialystok, The Medical University of Bialystok Clinical Hospital, Bialystok
  - Department of Cardiology and Structural Heart Diseases, Medical University of Silesia, Katowice, Poland, Katowice

IPD SHARING:
Plan to Share IPD: Undecided